CLINICAL TRIAL: NCT00398502
Title: A Randomized, Open-label, 3-period Crossover Study to Determine the Relative Bioavailability of Two Oral Formulations of MOA-728 and to Compare the Pharmacodynamics of the Two Oral Formulations of MOA-728 and the Subcutaneous Formulation in Subjects on Stable Methadone Maintenance
Brief Title: Comparisons Of The Bioavailability And Pharmacodynamics Of Various Formulations Of MOA-728 In Subjects On Methadone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Jeff Cohn, Salix Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3200A3-105
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Metahdone-maintenance Subjects

INTERVENTIONS:
Drug: MOA-728

SUMMARY:
Primary: To determine the relative bioavailability of MOA-728, an investigational drug, administered orally in both the capsule and tablet formulations to methadone maintenance subjects.Secondary: To assess the pharmacodynamic effect of MOA-728 administered both orally and subcutaneously to methadone maintenance subjects using the oral-cecal transit time.

ELIGIBILITY:
* Men or nonlactating and nonpregnant women, aged 18 to 65 years, inclusive. Women of nonchildbearing potential must be surgically sterile (hysterectomy, oophorectomy, and/or tubal ligation) or postmenopausal for ³1 year. Women of childbearing potential must be using an acceptable nonhormonal method of contraception (intrauterine device [IUD], diaphragm, or condom with spermicidal jelly or foam, or abstinence) for a period of at least 1 month before and after dose administration. All women must have negative pregnancy test results within 48 hours before the start of the first test article administration.
* Body mass index in the range of 18 to 35 kg/m² and body weight ≥50 kg.
* Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and 12-lead electrocardiogram (ECG).
* Subjects with positive results for HBsAg, and/or HCV antibodies may be enrolled if their bilirubin and serum albumin values are within normal limits and their liver function tests are within 1.2 times the upper limit of the normal range.
* A history of methadone treatment for at least 1 month before day -1 and have a positive drug test for methadone.
* No concomitant medication with the exception of stable doses of anxiolytic agents, antidepressants, Seroquel, occasional sleep medications, and drugs or supplements required to enhance or maintain regulation of bowel movements (must be stopped for the 72 hours before the first dose of test article administration in each period).
* Must have a high probability for compliance with and completion of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-10; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics and Pharmacodynamics

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Cohn, Study Director — Bausch Health Americas, Inc.
Locations (1):
- Gainesville, Florida, United States